CLINICAL TRIAL: NCT00387231
Title: Swiss Interventional Study on Silent Ischemia (SWISSI 2)
Brief Title: Comparison of Anti-Ischemic Drug Therapy and Percutaneous Transluminal Angioplasty After Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2006-10

CONDITIONS: Myocardial Ischemia
Keywords: Myocardial Ischemia; Randomized Controlled Trials; Angioplasty, Transluminal, Percutaneous Coronary; Drug Therapy
MeSH Terms: conditions — Myocardial Ischemia | interventions — Methods

INTERVENTIONS:
Procedure: Percutaneous coronary angioplasty/intervention (PCI)
Drug: Anti-ischemic drug therapy

SUMMARY:
Silent ischemia has been shown to negatively affect prognosis in patients after myocardial infarction. However, long-term outcome data in totally asymptomatic patients is missing and it is unknown whether angioplasty in addition to secondary preventive measures is superior to antiischemic drug therapy in these patients. Therefore, the SWISSI 2 study was started 15 years ago with the aim of comparing the effects of angioplasty with medical therapy on long-term outcome in patients with recent myocardial infarction and silent ischemia.

DETAILED DESCRIPTION:
Silent ischemia has been shown to negatively affect prognosis in patients after myocardial infarction (MI). Despite these consistent findings, there are almost no prospective data unequivocally documenting a benefit of antiischemic therapy on prognosis in patients with silent ischemia. There is some indirect evidence of a better outcome after repeat angioplasty for silent restenosis. In patients with a recent MI, the Asymptomatic Cardiac Ischemia Pilot study documented a short-term benefit of antiischemic drug therapy and angioplasty in patients with silent and symptomatic ischemic episodes. However, long-term outcome data in totally asymptomatic patients is missing and it is unknown whether angioplasty in addition to secondary preventive measures is superior to antiischemic drug therapy in these patients. Therefore, the (SWISSI 2) study was started 15 years ago with the aim of comparing the effects of angioplasty with medical therapy, each combined with secondary preventive advice, aspirin and statin therapy, on long-term outcome in patients with recent MI and an exercise test without symptoms but silent ischemia verified by stress imaging.

ELIGIBILITY:
Inclusion Criteria:

* Recent myocardial infarction within last 3 months
* Documented silent myocardial ischemia (type I)

Exclusion Criteria:

* Symptomatic myocardial ischemia

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-06; Study Completion 2006-05

PRIMARY OUTCOMES:
Combination of cardiac death, non-fatal myocardial infarction, and symptom-driven revascularization

SECONDARY OUTCOMES:
Overall mortality; Cardiac death; Non-fatal myocardial infarction; Symptom-driven revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Erne, MD, Study Chair — Department of Cardiology, Hospital Lucerne; Paul Erne, MD, Principal Investigator — Department of Cardiology, Hospital Lucerne
Locations (1):
- Department of Cardiology, Hospital Lucerne, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Derived] Schoenenberger AW, Jamshidi P, Kobza R, Zuber M, Stuck AE, Pfisterer M, Erne P. Progression of coronary artery disease during long-term follow-up of the Swiss Interventional Study on Silent Ischemia Type II (SWISSI II). Clin Cardiol. 2010 May;33(5):289-95. doi: 10.1002/clc.20775. PMID 20513067
- [Derived] Erne P, Schoenenberger AW, Burckhardt D, Zuber M, Kiowski W, Buser PT, Dubach P, Resink TJ, Pfisterer M. Effects of percutaneous coronary interventions in silent ischemia after myocardial infarction: the SWISSI II randomized controlled trial. JAMA. 2007 May 9;297(18):1985-91. doi: 10.1001/jama.297.18.1985. PMID 17488963